CLINICAL TRIAL: NCT00813683
Title: Study of Cephalic Version by Acupuncture for Breech Presentation.
Brief Title: Cephalic Version by Acupuncture for Breech Presentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3993
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breech Presentation
Keywords: Acupuncture, moxybustion,; Cephalic version,; Breech presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stimulation of "67 Bladder" point
  Interventions: Other: Acupuncture stimulation
- 2 (Sham Comparator): Stimulation of "45 Stomach" point (sham)
  Interventions: Other: Acupuncture stimulation

INTERVENTIONS:
Other: Acupuncture stimulation — Acupuncture by stimulation of "67 Bladder" point
  Arms: 1
Other: Acupuncture stimulation — Acupuncture stimulation of "45 Stomach" point (sham)
  Arms: 2

SUMMARY:
We want to study the efficiency of acupuncture for cephalic version of breech presentation during pregnancy.

Several randomized studies show that acupuncture may be useful in version of breech presentation, but none with a sham.

Protocol :

* Inclusion of patients with fetus in breech presentation at 32-34 weeks of pregnancy.
* Randomization. First group : acupuncture by stimulation of "67 Bladder" point.Second group : stimulation of "45 Stomach" point (sham).
* Ultrasonographic control of presentation at 35 weeks.

ELIGIBILITY:
Inclusion criteria:

* Single pregnancy at 32-34 weeks of pregnancy.
* Fetus in breech presentation.

Exclusion criteria:

* Twins.
* Story of preterm birth or any preterm birth risk
* Fetal malformations, abnormal karyotype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cephalic or breech presentation (ultrasonographic control at 35 weeks of pregnancy) | 35 weeks

SECONDARY OUTCOMES:
general outcomes about external cephalic version, delivery and neonates | 35 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Romain FAVRE, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Gynécologie-Obstétrique, Hôpital SIHCUS - CMCO, 19 rue Louis Pasteur, Schiltigheim, France

REFERENCES:
- [Result] Sananes N, Roth GE, Aissi GA, Meyer N, Bigler A, Bouschbacher JM, Helmlinger C, Viville B, Guilpain M, Gaudineau A, Akladios CY, Nisand I, Langer B, Vayssiere C, Favre R. Acupuncture version of breech presentation: a randomized sham-controlled single-blinded trial. Eur J Obstet Gynecol Reprod Biol. 2016 Sep;204:24-30. doi: 10.1016/j.ejogrb.2016.07.492. Epub 2016 Aug 2. PMID 27521594